CLINICAL TRIAL: NCT01567579
Title: An Evaluation of Routine Developmental Follow-Up in Infants and Children With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Cheryl Brosig, Professor, Pediatrics, Cardiology, Medical College of Wisconsin
Other Study IDs: CHW 09/98, GC 896
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Congenital Heart Defects
Keywords: congenital heart defects
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to understand how having a heart problem affects development,quality of life, and family life in young children and their families. Results for children and families with heart disease will be compared to children and families without heart disease. The investigators hope that this information may help us to support children and families better in the future. All children and families that are seen in the HHC Developmental Follow-Up Program will be asked if they would like to take part in this study. It is hypothesized that children with congenital heart disease will demonstrate developmental delays when compared to normative values.

DETAILED DESCRIPTION:
Research suggests that children with congenital heart disease are at higher risk for neurodevelopmental and psychosocial problems. Routine developmental screening and early intervention have been suggested as strategies to identify and ameliorate these problems. The purpose of this study is to describe the developmental trajectory and psychosocial functioning of children referred to the Herma Heart Center Developmental Follow-Up Program for routine developmental assessment.

The specific aims of this project are:

1. to summarize the results of developmental screening, quality of life, and family impact in subjects that have been evaluated in the HHC Developmental Follow-Up Program since its inception in 2007,
2. to evaluate longitudinal changes in the trajectory of development for subjects that undergo repeated developmental and psychosocial screening,
3. to characterize how subjects with congenital heart disease compare to normative data for the instruments utilized and samples of children with other chronic health conditions, and
4. to determine what factors predict variability in developmental outcomes i.e. demographic and clinical variables such as gender, race, socioeconomic status, diagnosis, type of surgery, and length of hospitalization among others.

Because our research and the research of others have indicated that children with Congenital Heart Disease (CHD) are at higher risk for neurodevelopmental and psychosocial problems, the Herma Heart Center Developmental Follow-Up Program was created in 2007. All infants who have open-heart surgery within the first 30 days of life, and all children under the age of 3 years who have a cyanotic lesion are referred to the clinic.

This study will utilize both retrospective chart review and prospective collection of data from new subjects entering the program.

No additional procedures are required to participate in the research study. Participation in the research study involves granting permission for the research team to systematically analyze the data obtained during the HHC Developmental Follow-Up Program clinic visits that a child participates in and to aggregate these data with all subjects that have received these follow-up assessments.

A sample size of 1000 subjects is needed to ensure adequate power to detect medium effect sizes for the multiple outcome measures that are proposed (assuming p = .05 and power = .80). Therefore, recruitment for the study will continue until a sample size of 1000 subjects is reached. Estimated recruitment duration is 7 years.

There are no anticipated risks related to participation in this study.

Descriptive analyses will be conducted to summarize characteristics of the sample and to determine the frequency of developmental/behavioral/emotional problems among children in the present sample. Correlation and regression analyses will be conducted to examine the relationships among demographic, clinical, and outcome variables. For children with multiple visits, longitudinal changes and the pattern of developmental trajectory for children with congenital heart disease will be examined.

Results may point to possible areas for intervention to improve child and family psychosocial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the Herma Heart Center (HHC)Developmental Follow-Up Clinic for assessment.

Exclusion Criteria:

* Non-English and Non-Spanish speaking families
* Children with extremely complex co-morbidities

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who have had congenital heart surgery, before the age of 1.
Sampling Method: Non-Probability Sample
Enrollment: 928 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Bayley Scales of Infant and Toddler Development Third Edition | every 6 months
  test of developmental skills

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L Brosig, PhD, Principal Investigator — Medical College of Wisconsin; Laurel M Bear, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Result] Soto CB, Olude O, Hoffmann RG, Bear L, Chin A, Dasgupta M, Mussatto K. Implementation of a routine developmental follow-up program for children with congenital heart disease: early results. Congenit Heart Dis. 2011 Sep-Oct;6(5):451-60. doi: 10.1111/j.1747-0803.2011.00546.x. Epub 2011 Jul 1. PMID 21718458
- [Result] Mussatto KA, Hoffmann RG, Hoffman GM, Tweddell JS, Bear L, Cao Y, Brosig C. Risk and prevalence of developmental delay in young children with congenital heart disease. Pediatrics. 2014 Mar;133(3):e570-7. doi: 10.1542/peds.2013-2309. Epub 2014 Feb 2. PMID 24488746
- [Result] Mussatto KA, Hoffmann R, Hoffman G, Tweddell JS, Bear L, Cao Y, Tanem J, Brosig C. Risk Factors for Abnormal Developmental Trajectories in Young Children With Congenital Heart Disease. Circulation. 2015 Aug 25;132(8):755-61. doi: 10.1161/CIRCULATIONAHA.114.014521. PMID 26304667
- [Result] Brosig CL, Bear L, Allen S, Hoffmann RG, Pan A, Frommelt M, Mussatto KA. Preschool Neurodevelopmental Outcomes in Children with Congenital Heart Disease. J Pediatr. 2017 Apr;183:80-86.e1. doi: 10.1016/j.jpeds.2016.12.044. Epub 2017 Jan 9. PMID 28081891
- [Result] Brosig CL, Bear L, Allen S, Simpson P, Zhang L, Frommelt M, Mussatto KA. Neurodevelopmental outcomes at 2 and 4 years in children with congenital heart disease. Congenit Heart Dis. 2018 Sep;13(5):700-705. doi: 10.1111/chd.12632. Epub 2018 Sep 6. PMID 30191663
- [Result] Jilek E, Shields A, Zhang L, Simpson P, Bear L, Martins SA, Mussatto KA, Brosig CL. Predictors of behavioural and emotional outcomes in toddlers with congenital heart disease. Cardiol Young. 2022 Aug;32(8):1216-1221. doi: 10.1017/S1047951121003942. Epub 2021 Sep 22. PMID 34548125